CLINICAL TRIAL: NCT06272461
Title: The Effect of Intravenous Lidocaine or Ketamine on Interleukin-6 Levels in Patients Undergoing Colorectal Surgery for Cancer: A Randomized Controlled Trial
Brief Title: Comparison of Intravenous Lidocaine vs Ketamine in Colorectal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, HibetAllah Ktata, Associate Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UTEM ELKI
Record Dates: First submitted 2024-01-19; First posted 2024-02-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Colorectal (Colon or Rectal) Cancer; Inflammation
MeSH Terms: conditions — Colonic Neoplasms; Inflammation

STUDY DESIGN:
Intervention Model Description: Intravenous Lidocaine vs intravenous ketamine
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV-Lido (Experimental): Intravenous Lidocaine dose loading than continuous infusion
  Interventions: Drug: Lidocaine IV
- IV-Keta (Active Comparator): Intravenous Ketamine dose loading than continuous infusion
  Interventions: Drug: Ketamine Injectable Solution

INTERVENTIONS:
Drug: Lidocaine IV — Intravenous Lidocaine Vs intravenous Ketamine in colorectal surgery for cancer
  Arms: IV-Lido
Drug: Ketamine Injectable Solution — Intravenous Lidocaine Vs intravenous Ketamine in colorectal surgery for cancer
  Arms: IV-Keta

SUMMARY:
Patients undergoing open colorectal surgery were randomly divided into two groups: Intravenous Lidocaine (IV-Lido) vs Intravenous Ketamine (IV-Keta).

For the IV-Lido group, patients received a loading dose of Lidocaine than a continuous infusion over twenty-four hours.

For the IV-Keta goup, patients received a loading dose of Ketamine than a continuous injection of Ketamine over twenty-four hours.

Plasma concentrations of Interleukin-6(IL-6) were measured preoperatively before anesthetic induction and at twenty-four hour post operatively.

DETAILED DESCRIPTION:
Patients undergoing open colorectal surgery with tumor resection were randomised prospectively into two groups: Intravenous Lidocaine (IV-Lido) vs Intravenous Ketamine (IV-Keta).

For the IV-Lido group (n=25), patients received a loading dose of 1.5 mg/kg of Lidocaine than a continuous infusion of 1.5 mg/kg/h over twenty-four hours.

For the IV-Keta goup(n=25), patients received a loading dose of 0.15mg/kg of Ketamine than a continuous injection of 0.15 mg/kg/h of Ketamine over twenty-four hours.

For both groups, plasma concentrations of Interleukin-6(IL-6) were measured preoperatively before anesthetic induction and at twenty-four hour post operatively. Plasma IL-6 concentrations at each point were compared between the groups.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients aged 18 or older.
* American society of anesthesiologists' (ASA) physical status of I-III.
* Elective open colorectal surgery.

NON INCLUSION CRITERIA:

* Patients with contraindications to lidocaine or ketamine.
* Corticosteroid therapy within the last 6 months.
* History of immunosuppressive therapy.
* History of surgery in the last 3 months.
* Personal medical history of inflammatory bowel disease.
* Personal medical history of cardiac arrythmias or conduction disorders.
* Alcohol or drug abuse.
* Chronic use of opioids or benzodiazepines.

EXCLUSION CRITERIA:

* Severe intraoperative complications.
* Duration of surgery longer than 5 hours.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
The variation of Interleukin-6 levels | 24 hours after surgery
  The difference of Interleukine-6 (IL-6) plasma concentration between baseline values and 24 hours after surgery.

SECONDARY OUTCOMES:
Pain assessed by Numerical Rating Scale (NRS) | Postoperatively, at Hour 2, Hour 12 and Hour 24. the patient asked to circle the number between 0 and 10:"0" usually represents 'no pain at all' whereas "10" represents 'the worst pain ever possible'.
  Postoperative pain was assessed by the Numerical Rating Scale (NRS)
Post-operative nausea and vomiting | During the first 24 hours postoperatively
  Incidence of post-operative nausea and vomiting during the first 24 hours.
Bowel function. | During the first 24 hours postoperatively
  Time to return of bowel function.
Hospital length of stay. | From date of randomization until the date of to discharge from the hospital assessed up to 15 days
  Hospital length of stay ( in days)
Post-operative complications. | From date of randomization until the date of to discharge from the hospital assessed up to 15 days
  Incidence of intrahospital post-operative complications.

CONTACTS AND LOCATIONS:
Overall Officials: BEN ALI MECHAAL, Professor, Principal Investigator — university manar Tunis, Tunisia
Locations (1):
- Tunisia, Nabeul, Tunisia